CLINICAL TRIAL: NCT02610582
Title: Safety and Efficacy of a Bilateral Single Subretinal Injection of rAAV.hCNGA3 in Adult and Minor Patients With CNGA3-linked Achromatopsia Investigated in a Randomized, Wait List Controlled, Observer-masked Trial
Brief Title: Safety and Efficacy of rAAV.hCNGA3 Gene Therapy in Patients With CNGA3-linked Achromatopsia
Acronym: Colourbridge
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: STZ eyetrial (Other)
Collaborators: University Hospital Tuebingen (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RDC-CNGA3-01; 2014-001874-32 (EudraCT Number); 096/2015 AMG1 (Other: Ethics Committee Tübingen)
Record Dates: First submitted 2015-09-18; First posted 2015-11-20 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Achromatopsia
Keywords: CNGA3-linked
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment arm (Other): single subretinal injection of 1x10e11 vector genome particles of rAAV.hCNGA3 in each eye at different time-points
  Interventions: Drug: rAAV.hCNGA3
- Waiting group Arm (Other): Waiting group will serve as comparator group first and will receive the treatment at a later timepoint.
  Interventions: Drug: rAAV.hCNGA3

INTERVENTIONS:
Drug: rAAV.hCNGA3 — Single subretinal injection of rAAV.hCNGA3

SUMMARY:
The purpose of this study is to proof the safety and efficacy of a single bilateral subretinal injection of rAAV.hCNGA3 in adult and minor patients with CNGA3-linked achromatopsia.

DETAILED DESCRIPTION:
Title: Safety and efficacy of a bilateral single subretinal injection of rAAV.hCNGA3 in adult and minor patients with CNGA3-linked achromatopsia investigated in a randomized, wait list controlled, observer-masked trial

Phase: I/II

Indication: CNGA3-linked achromatopsia

Aim: to proof the safety and efficacy of a single bilateral subretinal injection of rAAV.hCNGA3 in adult and minor patients with CNGA3-linked achromatopsia.

Study design: open, mono-center, randomized, wait list controlled, observer-masked trial

Study Population:

Inclusion Criteria (Both Eyes)

* clinical diagnosis of achromatopsia
* 6-12 years of age
* ≥ 18 years of age
* confirmed mutation in CNGA3
* BCVA ≥ 20/400
* a minimal outer nuclear layer thickness of 10µm at 3° eccentricity (normal = 38±6µm)
* ability to understand and willingness to consent to study protocol
* no infection with Human Immundeficiency Virus (HIV)
* Male patients must agree to use condoms during the first 6 months post treatment.
* Female patients of childbearing potential must agree to use an effective method of birth control during the first 6 months post treatment.
* negative pregnancy test in women with childbearing potential (a woman who is two years post-menopausal or surgically sterile is not considered to be of childbearing potential)

Exclusion Criteria

* • any other retinopathy due to other diseases e.g. (but not limited to) arterial hypertension, trauma or acquired inflammatory diseases (uveitis serology) , retinopathy of the premature
* systemic conditions (e.g. coronary heart disease, congenital/genetic conditions, autoimmune disorders) which may affect study participation or outcome measures
* current or recent participation in other study or administration of biologic agent within the last three months
* recent (6 months) ocular surgery, intravitreal or subretinal implantation of a medical device
* known sensitivity to any compound used in the study
* contraindications to systemic immunosuppression
* subject/partner of childbearing potential unwilling to use adequate contraception for six months after dosing
* nursing or pregnant female subject women
* any other cause that, in the investigator's opinion, renders potential subjects not suitable for the study
* mutations in another achromatopsia gene
* contraindications in view of the planned surgery (e.g. anaemia Hb<8g/dl, severe coagulopathy, severe blood pressure fluctuations) including intolerance and contraindications to general anaesthesia
* ocular opacity and mature cataract
* ocular infection with herpes simplex virus in medical history
* history of ocular malignancies
* disorders of the internal retina (e.g. retinal detachment in the patients history)
* glaucoma defined as damage of the optic nerve
* vascular retinal occlusion
* history of poorly controlled (HbA1c > 7%) Diabetes Mellitus type 1 or type 2
* patients treated with systemic corticoids within 14 days prior inclusion
* systemic illness or medically significant abnormal laboratory values >3 UNL in blood analysis including renal and hepatic functions at inclusion
* absence of vision on the other contralateral eye
* contraindication to pharmacological mydriasis (e.g. history of angle block glaucoma)

Patient Number: 3 Strata: Cohort A n = 4, ≥ 18 years of age and previous participation in phaseI/II, Cohort B n = 4, ≥ 18 years of age, Cohort C n= 6, 6-12 years of age

Treatment:

Each cohort will receive a single subretinal injection of 1x10e11 vector genome particles of rAAV.hCNGA3 in each eye at different time-points. Cohort A, in whom the first eye has received treatment under protocol version 5.0, will only receive one injection in the second eye.

After standard three-port 23G pars plana vitrectomy, balanced salt solution will be used to induce a localized primary retinal detachment in a controlled fashion. Vector solution will be applied using disposable 41G extendible subretinal injection needles within a standard 23G body to fit the port system.

Primary Endpoint:

Primary endpoint safety: Safety assessment 12 months after treatment, descriptively Primary endpoint efficacy: Contrast sensitivity (Pelli Robson 3 m) 6 months after treatment

Key secondary endpoints efficacy 12 months after treatment:

* Contrast sensitivity (Pelli Robson 3 m)
* BCVA assessed using the ETDRS visual acuity protocol
* Microperimetry (MAIA) (20°)
* Chromatic Pupil Campimetry
* Patient reported outcomes (VFQ25/CVFQ, A3-PRO) Safety as the primary endpoint will be assessed by clinical examination of ocular inflammation (slit lamp, fundus biomicroscopy, fundus photography. Systemic safety will be assessed by vital signs, routine clinical chemistry testing (including CRP, ESR) and full/differential blood counts. Immunopathology essays will include specific enzyme-linked immunosorbent assays for humoral antibodies against rAAV8 capsid protein. Biodistribution will be monitored by polymerase chain reaction studies on rAAV8 genome in blood, urine, saliva and tear fluid.

Statistical Methods:

Efficacy: The analysis of the primary endpoint (contrast sensitivity after 6 months) will be done using a pre / post comparison for the entire sample including both eyes for cohort B and C (n=10) and only one eye for cohort A (n=4) with GEE correction for the dependency of left and right eye. In the waiting group the second (therapeutic) phase will be used. The dependency appears for cohorts B and C which contribute both eyes but not for cohort A which contributes only one eye to the efficacy analysis. The study is powered for this analysis. We will use the specific type of IEE (Independence Estimating Equations) which reveals correct standard errors and a robust estimate for model parameters.

Additionally, we will compare the Intervention group vs. control group (waiting group) (n=7 vs. 7), using baseline adjusted analysis of covariance and between subject comparisons. This analysis will use GEEs as described for the primary analysis including both eyes of cohort B and C and only the newly treated eye in cohort A. This analysis will be descriptive and provide evidence for the planning of a randomized Phase III trial.

The primary analysis population will be the ITT in which only patients with baseline measurements will be included. For patients providing baseline measurements in one eye, only this eye will be included. Multiple imputation will be done with sampling unit "eye" if only baseline, but not follow up data are available. Descriptive parameters will be given for the full cohort (n=14) and for the sub-strata (n=4, 4, 6 pooled), additionally, correlation analysis descriptively for the comparison of subjective and objective measurements will be done.

Safety (ITT): AEs and SAEs will be documented using line listings and tabulations (MedDRA code will be applied). Frequency tabulations of certain classes of events will be given including two-sided 95% confidence intervals.

The aim of analysis (1) is to gain evidence for a sample size estimation for a phase III trial with similar design, where analysis (2) will be confirmatory and powered according to a sample size estimation.

Time Schedule: of trial November 2015 end of recruitment 04/2022, end of trial 04/2027, duration of trial per patient: one year with four years of follow-up.

The final study report will be prepared after completion of the four year follow-up period (5 years after treatment).

ELIGIBILITY:
Inclusion Criteria (Both Eyes)

* clinical diagnosis of achromatopsia
* 6-12 years of age
* ≥ 18 years of age
* confirmed mutation in CNGA3
* BCVA ≥ 20/400
* a minimal outer nuclear layer thickness of 10µm at 3° eccentricity (normal = 38±6µm)
* ability to understand and willingness to consent to study protocol
* no infection with Human Immundeficiency Virus (HIV)
* Male patients must agree to use condoms during the first 6 months post treatment.
* Female patients of childbearing potential must agree to use an effective method of birth control during the first 6 months post treatment.
* negative pregnancy test in women with childbearing potential (a woman who is two years post-menopausal or surgically sterile is not considered to be of childbearing potential)

Exclusion Criteria

* any other retinopathy due to other diseases e.g. (but not limited to) arterial hypertension, trauma or acquired inflammatory diseases (uveitis serology) , retinopathy of the premature
* systemic conditions (e.g. coronary heart disease, congenital/genetic conditions, autoimmune disorders) which may affect study participation or outcome measures
* current or recent participation in other study or administration of biologic agent within the last three months
* recent (6 months) ocular surgery, intravitreal or subretinal implantation of a medical device
* known sensitivity to any compound used in the study
* contraindications to systemic immunosuppression
* subject/partner of childbearing potential unwilling to use adequate contraception for six months after dosing
* nursing or pregnant female subject women
* any other cause that, in the investigator's opinion, renders potential subjects not suitable for the study
* mutations in another achromatopsia gene
* contraindications in view of the planned surgery (e.g. anaemia Hb<8g/dl, severe coagulopathy, severe blood pressure fluctuations) including intolerance and contraindications to general anaesthesia
* ocular opacity and mature cataract
* ocular infection with herpes simplex virus in medical history
* history of ocular malignancies
* disorders of the internal retina (e.g. retinal detachment in the patients history)
* glaucoma defined as damage of the optic nerve
* vascular retinal occlusion
* history of poorly controlled (HbA1c > 7%) Diabetes Mellitus type 1 or type 2
* patients treated with systemic corticoids within 14 days prior inclusion
* systemic illness or medically significant abnormal laboratory values >3 UNL in blood analysis including renal and hepatic functions at inclusion
* absence of vision on the other contralateral eye
* contraindication to pharmacological mydriasis (e.g. history of angle block glaucoma)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety (AE). Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | Day 0 - Day 365
  Safety as the primary endpoint will be assessed by clinical examination of ocular inflammation (slit lamp, fundus biomicroscopy, fundus photography. Systemic safety will be assessed by vital signs, routine clinical chemistry testing (including CRP, ESR) and full/differential blood counts. Immunopathology essays will include specific enzyme-linked immunosorbent assays for humoral antibodies against rAAV8 capsid protein. Biodistribution will be monitored by polymerase chain reaction studies on rAAV8 genome in blood, urine, saliva and tear fluid.

SECONDARY OUTCOMES:
Efficacy measures. Number of Participants With improved Visual Function. | Day 14 - Day 365
  The investigation of treatment effects as reflected by patient/parent reported outcomes and the efficacy of the intervention on visual function, as well as the evaluation of retinal imaging (safety) are secondary aims of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Fischer, Prof., Principal Investigator — University Hospital Tuebingen, Center for Ophthalmology
Locations (1):
- University Hospital Tuebingen, Center for Ophthalmology, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reichel FF, Michalakis S, Wilhelm B, Zobor D, Muehlfriedel R, Kohl S, Weisschuh N, Sothilingam V, Kuehlewein L, Kahle N, Seitz I, Paquet-Durand F, Tsang SH, Martus P, Peters T, Seeliger M, Bartz-Schmidt KU, Ueffing M, Zrenner E, Biel M, Wissinger B, Fischer D. Three-year results of phase I retinal gene therapy trial for CNGA3-mutated achromatopsia: results of a non randomised controlled trial. Br J Ophthalmol. 2022 Nov;106(11):1567-1572. doi: 10.1136/bjophthalmol-2021-319067. Epub 2021 May 18. PMID 34006508
- [Derived] Fischer MD, Michalakis S, Wilhelm B, Zobor D, Muehlfriedel R, Kohl S, Weisschuh N, Ochakovski GA, Klein R, Schoen C, Sothilingam V, Garcia-Garrido M, Kuehlewein L, Kahle N, Werner A, Dauletbekov D, Paquet-Durand F, Tsang S, Martus P, Peters T, Seeliger M, Bartz-Schmidt KU, Ueffing M, Zrenner E, Biel M, Wissinger B. Safety and Vision Outcomes of Subretinal Gene Therapy Targeting Cone Photoreceptors in Achromatopsia: A Nonrandomized Controlled Trial. JAMA Ophthalmol. 2020 Jun 1;138(6):643-651. doi: 10.1001/jamaophthalmol.2020.1032. PMID 32352493